CLINICAL TRIAL: NCT04729842
Title: Comparison Between Bupivacaine and Ropivacaine in Patients Undergoing Forearm Surgeries Under Axillary Brachial Plexus Block: A Prospective Comparative Randomized Study
Brief Title: Comparison Between Bupivacaine and Ropivacaine in Patients Undergoing Forearm Surgeries Under Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assam Medical College (Other)
Responsible Party: Principal Investigator, Dr Karuna Kumar Das, Associate Professor, Department of Anaesthesiology and Critical care, Assam Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AssamMC
Record Dates: First submitted 2021-01-21; First posted 2021-01-29 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: a prospective randomized single-blind study. Patients were blind to the study of drugs. Blinding was achieved by the examiner of the study. Participants were randomly allocated into two groups (Group - B i.e. Bupivacaine Group and Group - R i.e. Ropivacaine group) using computer-generated randomization and allocation concealment was done using sealed sequentially numbered containers opaque envelope technique (SNOSE)
Who Masked: Participant
Masking Description: Patients were blind to the study of drugs. Blinding was achieved by the examiner of the study. The allocation concealment was done using sealed sequentially numbered containers opaque envelope technique and the identical-looking container was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group - B , Patients who recieved Bupivacaine (Active Comparator): 30 ml of 0.5% bupivacaine was injected equally divided and injected in four nerves (musculocutaneous, median, radial and ulnar nerves)
  Interventions: Procedure: Axillary Brachial plexus block
- Group - R , Patients who received Ropivacaine (Active Comparator): 30 ml of a solution containing 0.5% ropivacaine was equally divided and injected in the four nerves (musculocutaneous, median, radial and ulnar nerves)
  Interventions: Procedure: Axillary Brachial plexus block

INTERVENTIONS:
Procedure: Axillary Brachial plexus block — Brachial plexus block via axillary route was administered using 30 ml of 0.5% Bupivacaine in group B and 30 ml of 0.5% Ropivacaine in Group R
  Other Names: Brachial plexus block for forearm surgeries

SUMMARY:
This prospective comparative randomized study was done to compare Bupivacaine and Ropivacaine in patients undergoing forearm surgeries under axillary brachial plexus block. The study compares the onset and duration of sensory block, onset and duration of motor block and duration of analgesia between these two drugs.

DETAILED DESCRIPTION:
This is a prospective comparative randomized study to compare Bupivacaine and Ropivacaine in patients undergoing forearm surgeries under axillary brachial plexus block. A sample size of 100 was considered who are meeting the inclusion and exclusion criteria were selected, and divided into two groups of 50 each using computer-generated randomization and allocation concealment was done using sealed sequentially numbered containers opaque envelope technique (SNOSE). One group will receive Bupivacaine and the other Ropivacaine. Patients were blind to the study. In the Bupivacaine group, 30 ml of 0.5% bupivacaine was injected equally divided and injected in four nerves (musculocutaneous, median, radial and ulnar nerves). In the Ropivacaine group, 30 ml of a solution containing 0.5% ropivacaine was equally divided and injected in the four nerves. Sensory block was tested with a 22-gauge hypodermic needle by using the pinprick test and compared with the contralateral hand. Sensory block was graded as Grade 0: Sharp pin felt, Grade 1: Analgesia, dull sensation felt and Grade 2: Anaesthesia, no sensation felt. Motor function was assessed as per the modified Bromage scale. 0: Able to raise the extended arm to 90 degrees for a full 2 sec, 1: Able to flex the elbow and move the fingers but unable to raise the extended arm, 2: Unable to flex the elbow but able to move the fingers and 3: Unable to move the arm, elbow or fingers. The onset of sensory blockade was assessed by the time from the completion of injection of the study drug till the loss of pinprick sensation. It was assessed every minute. The onset of motor blockade was assessed when there was Grade 1 motor blockade. It was assessed every minute. Duration of sensory blockade was assessed by the time between onset of sensory blockade and return of dull sensation to pinprick. .It was assessed every 15 minutes. Duration of motor blockade was assessed by the time between onset of motor blockade and time at which patients could first move their fingers. It was assessed every 15minutes. Duration of analgesia is the time interval between the onset of sensory block and the patient's first analgesic request. The rescue analgesia in the form of inj. Diclofenac sodium (1.5 mg/kg) intramuscularly was given. Block was considered to have failed when sensory anaesthesia was not achieved within 30 min. General anaesthesia was given subsequently to these patients and was excluded from the study. Again, a patient showing an allergic reaction to the intervention were also withdrawn from the study.

Statistical Analysis - Normally distributed quantitative data were presented as mean ± SD, whereas data not normally distributed were presented as median (IQR). While comparing quantitative data between the two groups, for normally distributed quantitative data, Independent student t-test was used, on the other hand, Mann-Whitney test was used. For comparing qualitative variable chi-square or Fischer exact test was applied as appropriate. In case of repeated measure data, mixed effect ANOVA was used. For all test P value of < 0.05 was considered as significant and P-value < 0.001 was considered as highly significant. SPSS version 21 (IBM, Newyork) was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients with ASA classes I and II who gave consent and were candidates for elective forearm surgeries.

Exclusion Criteria:

1. Any allergic reactions to ropivacaine, bupivacaine and lignocaine.
2. All patients with hypertension, cardiac, hepatic or renal diseases.
3. Pregnant women, drug abusers and psychiatric patients.
4. Patient who had an anatomical or vascular abnormality in the upper extremity.
5. Bleeding diathesis.
6. Local infection of the axilla.
7. Patient refusal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Onset of sensory block | Time in minutes from the completion of injection of the study drug till the loss of pinprick sensation. The estimated time frame from injection of study drug to onset of sensory block is 15 minutes.
  Sensory block was tested with a 22-gauge hypodermic needle by using the pinprick test and compared with the contra-lateral hand. Sensory block was graded as Grade 0: Sharp pin felt, Grade 1: Analgesia, dull sensation felt and Grade 2: Anaesthesia, no sensation felt.
Duration of sensory block | Time in minutes between onset of sensory blockade and return of dull sensation to pin prick. The estimated time frame for duration of sensory block is 540 minutes.
  Duration was assessed from loss of pinprick sensation to return of sensation.

SECONDARY OUTCOMES:
Onset of motor block | Time from the completion of injection of the study drug till the patient is unable to move his fingers. The estimated time frame for onset of motor block is 20 minutes.
  Motor function was assessed as per modified Bromage Scale . 0: Able to raise the extended arm to 90o for a full 2 sec, 1: Able to flex the elbow and move the fingers but unable to raise the extended arm, 2: Unable to flex the elbow but able to move the fingers and 3: Unable to move the arm, elbow or fingers .
Duration of motor block | Time in minutes between onset of motor blockade and time at which patient could first move their fingers. The estimated time frame for duration of motor block is 480 minutes.
  Duration was assessed from loss of motor function till the return of the function.
Duration of analgesia | Time in minutes between onset of sensory block and patient's first analgesic request. Time frame for duration of analgesia is 600 minutes
  Duration was assessed from the onset of loss of sensory function till the patient feels pain. The rescue analgesia in the form of inj. Diclofenac sodium (1.5 mg/kg) intramuscularly was given.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennan F, Lohman D, Gwyther L. Access to Pain Management as a Human Right. Am J Public Health. 2019 Jan;109(1):61-65. doi: 10.2105/AJPH.2018.304743. PMID 32941757
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Background] Armstrong KP, Cherry RA. Brachial plexus anesthesia compared to general anesthesia when a block room is available. Can J Anaesth. 2004 Jan;51(1):41-4. doi: 10.1007/BF03018545. PMID 14709459
- [Background] Clarkson CW, Hondeghem LM. Mechanism for bupivacaine depression of cardiac conduction: fast block of sodium channels during the action potential with slow recovery from block during diastole. Anesthesiology. 1985 Apr;62(4):396-405. PMID 2580463
- [Background] Hickey R, Hoffman J, Ramamurthy S. A comparison of ropivacaine 0.5% and bupivacaine 0.5% for brachial plexus block. Anesthesiology. 1991 Apr;74(4):639-42. doi: 10.1097/00000542-199104000-00002. PMID 2008942
- [Background] De Andres J, Sala-Blanch X. Peripheral nerve stimulation in the practice of brachial plexus anesthesia: a review. Reg Anesth Pain Med. 2001 Sep-Oct;26(5):478-83. doi: 10.1053/rapm.2001.26485. No abstract available. PMID 11561271
- [Background] Schulz KF, Grimes DA. Allocation concealment in randomised trials: defending against deciphering. Lancet. 2002 Feb 16;359(9306):614-8. doi: 10.1016/S0140-6736(02)07750-4. PMID 11867132
- [Background] Cline E, Franz D, Polley RD, Maye J, Burkard J, Pellegrini J. Analgesia and effectiveness of levobupivacaine compared with ropivacaine in patients undergoing an axillary brachial plexus block. AANA J. 2004 Oct;72(5):339-45. PMID 15529729
- [Background] Thornton KL, Sacks MD, Hall R, Bingham R. Comparison of 0.2% ropivacaine and 0.25% bupivacaine for axillary brachial plexus blocks in paediatric hand surgery. Paediatr Anaesth. 2003 Jun;13(5):409-12. doi: 10.1046/j.1460-9592.2003.01065.x. PMID 12791114
- [Background] Kooloth RA, Patel SN, Mehta MK. A comparison of 0.5% Ropivacaine and 0.5% Bupivacaine in supraclavicular brachial plexus block -. National Journal of Medical Research. 2015;5(1):67-70.
- [Result] Kaur A, Singh RB, Tripathi RK, Choubey S. Comparision between bupivacaine and ropivacaine in patients undergoing forearm surgeries under axillary brachial plexus block: a prospective randomized study. J Clin Diagn Res. 2015 Jan;9(1):UC01-6. doi: 10.7860/JCDR/2015/10556.5446. Epub 2015 Jan 1. PMID 25738062
- [Result] Rathod H, Parikh H, Upadhayaya RM. Comparative study of 0.375% bupivacaine and 0.375% ropivacaine in brachial plexus block via supraclavicular approach. Int Jour of Biomed Res. 2015 Feb 28;6(2):77-82.
- [Result] Modak S, Basantwani S. Comparative study of 0.5% ropivacaine and 0.5% bupivacaine for brachial plexus block by supraclavicular approach for upper limb surgeries. International Journal of Basic & Clinical Pharmacology. 2017 Jan 5;5(4):1205-9.
- See also: OpenEpi - Toolkit Shell for Developing New Applications [Internet]. — http://www.openepi.com/SampleSize/SSMean.htm